CLINICAL TRIAL: NCT04063319
Title: Nursing Students' Recognition of and Response to Deteriorating Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Agder (Other)
Responsible Party: Principal Investigator, Eli Andås, Senior Adviser, University of Agder
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 52110
Record Dates: First submitted 2019-06-21; First posted 2019-08-21 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Knowledge, Attitudes, Practice
Keywords: High-fidelity simulation; Self-confidence; Deteriorating patients; Ordinal data; Questionnaire
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-fidelity simulation (Experimental): The participants in the intervention group will receive an high-fidelity simulation intervention
  Interventions: Other: High-fidelity simulation
- Control (No Intervention): The participants in the control group will not receive any instructional intervention

INTERVENTIONS:
Other: High-fidelity simulation — The set up in the high-fidelity simulation intervention is a deteriorating patient scenario.
  Arms: High-fidelity simulation

SUMMARY:
The overall aim of this intervention study is to examine the effects of an high-fidelity simulation intervention in undergraduate nursing education developed to identify recognizing and responding to patient deterioration. Half of the participants will receive an intervention with high-fidelity simulation, while the other half will not receive any instructional intervention.

DETAILED DESCRIPTION:
Simulation-based nursing education is an increasingly used pedagogical approach.

The overall aim of this intervention study is to examine the effects of an high-fidelity simulation intervention developed to identify how recognizing and responding to patient deterioration improves the knowledge and self-confidence of undergraduate nursing students.

Specific aims:

1. To describe and estimate the change in undergraduate nursing students' knowledge and perceived self-confidence after an high-fidelity simulation intervention.
2. To identify the barriers and enablers that may impact on a successful implementation of the high-fidelity simulation intervention.

Half of the participants will receive an intervention with high-fidelity simulation, while the other half will not receive any instructional intervention. All participants will answer a questionnaire developed to measure perceived knowledge and levels of self-confidence pre- and post-intervention or before and after a meeting (control group). Five students and six faculty members will also be interviewed as a part of a process evaluation.

The study is part of a PhD project.

ELIGIBILITY:
Inclusion Criteria:

* All undergraduate nursing students at two universities enrolling in a specific course that includes high-fidelity simulation

Exclusion Criteria:

- None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2016-08-15 (Actual); Primary Completion 2018-12-16 (Actual); Study Completion 2018-12-16 (Actual)

PRIMARY OUTCOMES:
Knowledge | Baseline (immediately before intervention) and immediately after intervention (the intervention will last for 3 hours)
  Change in total score from 0-20 using 20 multiple choice questions about vital signs, clinical changes in vital signs after major acute blood loss, and nursing procedures. Higher scores at post-intervention represent a better outcome.

SECONDARY OUTCOMES:
Levels of self-confidence | Baseline (immediately before intervention) and immediately after intervention (the intervention will last for 3 hours)
  Change in total responses using 20 questions with five response alternatives (from not at all confident to very confident) about vital signs, clinical changes in vital signs after major acute blood loss, and nursing procedures . Higher scores at post-intervention represent a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Mariann Fossum, Professor, Study Chair — University of Agder

REFERENCES:
- [Derived] Haddeland K, Slettebo A, Fossum M. Enablers of the successful implementation of simulation exercises: a qualitative study among nurse teachers in undergraduate nursing education. BMC Nurs. 2021 Nov 22;20(1):234. doi: 10.1186/s12912-021-00756-3. PMID 34802428